CLINICAL TRIAL: NCT05023018
Title: An Open-Label, Phase 2 Study of NEO100 in Participants With Residual, Progressive or Recurrent High-Grade Meningioma
Brief Title: NEO100 and High-Grade Meningioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neonc Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO100-02
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Residual, Progressive or Recurrent Grade II or III Meningioma
Keywords: Residual, Progressive or Recurrent Grade II or III Meningioma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — perillyl alcohol

STUDY DESIGN:
Intervention Model Description: This multi-site, Phase 2 clinical trial is an open label study to identify the safety, pharmacokinetics, and efficacy of a repeated dose regimen of NEO100 (perillyl alcohol) for the treatment of patients with radiographically-confirmed residual, progressive or recurrent high-grade meningioma. There will be up to 30 patients enrolled into the study to enroll 28 evaluable patients. NEO100 will be self-administered four times daily for a 28-day treatment cycle until disease progression, death or patient withdraw for any reason, whichever occurs first.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with high-grade meningioma (Experimental): 30 patients with residual high-grade meningioma following resection surgery, radiographically-confirmed progression of high-grade meningioma or recurrent high-grade meningioma
  Interventions: Drug: NEO100

INTERVENTIONS:
Drug: NEO100 — NEO100 is a purified form of perillyl alcohol.

SUMMARY:
This multi-site, Phase 2 clinical trial is an open-label study to identify the safety, pharmacokinetics, and efficacy of a repeated dose regimen of NEO100 (perillyl alcohol) for the treatment of patients with residual high-grade meningioma following resection surgery, radiographically-confirmed progression of high-grade meningioma or recurrent high-grade meningioma. There will be up to 30 patients enrolled in this study to have 29 evaluable patients. NEO100 will be self-administered four times daily on a 28-day treatment cycle until disease progression, death or patient withdraw from study for any reason, whichever occurs first.

DETAILED DESCRIPTION:
Meningiomas are the most common primary brain tumor with an incidence rate of 8.33 per 100,000. They originate from the meningeal (dural) coverings of the brain and spinal cord. Although the majority of meningiomas are benign, these tumors can grow slowly until they are very large, if left undiscovered, and, in some locations can be severely disabling and/or life-threatening.

There is a relative paucity of prospective clinical trials that provide an evidenced-based agreed upon approach to managing meningioma. Furthermore, uniformly applied guidelines have been difficult to achieve given the typical pattern of slow growth.

Meningiomas can be organized into two groups. WHO Grade I meningioma are histologically benign and can be managed by careful observation as recommended in the National Comprehensive Cancer Network Guidelines. Grade I meningiomas are low grade and have a 7-20% recurrence risk. For most other patients (WHO Grade II and WHO Grade III) there is an increased risk of recurrence and death. Grade II meningiomas occur in 5-15% of cases with a 30-40% recurrence risk and Grade III meningiomas occur 1-3% of the time with a 50-80% recurrence risk. For Grade I and Grade II meningiomas, gross total resection is standard. WHO Grade II and WHO Grade III meningiomas are referred to as high-grade meningiomas.

Questions remain regarding the selection and timing of treatment, especially in cases of recurrent meningioma or newly diagnosed high-grade meningioma (WHO Grade II or Grade III meningioma). For patients undergoing definitive therapy, complete resection (gross total resection) has been the standard. However, there is a significant subset of patients who are not successfully managed by surgery alone, or in whom a complete resection is not possible due to the relationship of the tumor to important anatomy. Complete tumor resection is not always achievable as many meningiomas arise at or near critical neural or vascular structures or in sites with limited surgical access When a gross total resection cannot be accomplished, post-operative radiation therapy is often considered (e.g., single-session stereotactic radiosurgery, hypofractionated stereotactic radiation therapy and conventionally fractionated external beam radiation therapy).

The potential for recurrence, whether following subtotal resection or gross-total resection, is well recognized. As a result, there is increasing evidence from retrospective review of case histories in support of radiation therapy as primary therapy for high-grade meningioma (or radiation prior to or following resection surgery). The relative efficacy of these approaches has not yet been tested in rigorously designed prospective clinical trials.

The role of chemotherapy in treating meningioma is also unclear; however, there is a need for additional therapeutic options to treat meningioma cases which cannot be managed by surgery and/or radiation therapy alone.

One reason for the hesitation to treat primary central nervous system tumours with chemotherapy is the difficulty of penetrating the blood brain barrier with chemotherapy agents. Nasal brain delivery of chemotherapy offers a novel, paradigm shifting platform based on technology to deliver chemotherapy via inhalation to the brain tumor. The presumed mechanism of nasal brain delivery from preclinical rodent studies is thought to be via the olfactory and trigeminal nerves. Effective nasal brain delivery has been demonstrated in humans in other diseases. For example, Reger et al. have reported effective delivery of intranasal insulin for Alzheimer's disease.

Perillyl alcohol, also called p-metha1,7-diene-6-ol,or 4-isopropenylcyclo-hexenecarbinol, is a monoterpene, isolated from the essential oils of lavender, peppermint, spearmint, and several other plants and synthesized by the mevalonate pathway. It has been previously demonstrated to have anti-cancer properties in preclinical studies in rodent models for a variety of cancers including mammary, pancreatic, and colon cancer. Although the exact mechanism of perillyl alcohol induced tumor regression is unknown, perillyl alcohol has been reported to modulate cellular processes that control cell growth and differentiation including G1 cell cycle arrest and induction of apoptosis.

Perillyl alcohol has also been shown to inhibit post-translational modification of proteins involved in signal transduction. It has been postulated that the anti-neoplastic activity of perillyl alcohol involves a decrease in the levels of isoprenylated Ras and Ras-related proteins, thereby reducing the physiological functioning of these proteins. Protein isoprenylation involves the post-translational modification of a protein by the covalent attachment of a lipophilic farnesyl isoprenoid group to a cysteine residue at or near the carboxyl terminus. Isoprenoid substrates for prenylprotein transferase enzymes include farnesyl pyrophosphate plus geranylgeranyl pyrophosphate, two intermediates in the mevalonate pathway. This action was attributed to the inhibition of farnesyl protein transferase activity. Farnesylation is the most critical part of the process that leads to the activation of Ras, and farnesyl transferase inhibitors exert their antitumor effect in part by inhibiting Ras-mediated signaling. A study revealed that H-Ras and K-Ras farnesylation were inhibited by perillyl alcohol.

Ras activity is elevated in malignant central nervous system tumors. Strong evidence demonstrates that Ras protein is highly expressed in meningioma cells, and inhibition of Ras activity may inhibit the growth of meningiomas. Activated Ras stimulates other pathways essential for proliferation and progression through the cell cycle and inhibition of apoptosis in malignant gliomas. Moreover, the formation of malignant meningioma may require the cooperation of both Ras and Akt signaling. This cooperative effect has been demonstrated by somatic-cell gene transfer, during which transfer of either an activated form of K-Ras or Akt alone to neural progenitors was insufficient to form malignant glioma in vivo, but the combined effect of both pathways could initiate gliomagenesis. Thus, based on this potential alteration in signal transduction involving K-Ras in malignant central nervous system tumors, and its ability to induce cell cycle arrest and apoptosis, perillyl alcohol (NEO100) may be an attractive agent and warrants further clinical development. Furthermore, intranasal delivery of NEO100 has the additional, potential benefit of direct drug delivery into the brain and avoiding systemic toxicity and first pass metabolism.

Intranasal delivery of NEO100 will directly penetrate meningiomas, particularly skull-based meningiomas which extend along the olfactory groove, tuberculum sella, spenoid ridge and petroclival region. These represent some of the most challenging pathologies encountered by neurosurgeons due to the meningioma depth, invasion, vascularity and relationship to critical cranial nerves and vessels.

Intranasal perillyl alcohol has been tested in a Phase I clinical trial in the US, it has also been studied in two clinical studies in Brazil in more than 275 patients with systemic cancers and in malignant glioma. The Brazil studies indicate good tolerance and no long term central nervous system (CNS) or systemic severe adverse events. Adult patients with CNS cancers received commercial (Sigma Chemical) perillyl alcohol (formulated as a 10% solution in ethanol:glycerol) administered intranasally via a commercial nasal delivery mask four times a day (110 mg/dose or 440 mg/day). Radiographic regression and a PFS-6 of 50% were reported. A pharmacokinetic study showed that perillic acid, a metabolite of perillyl alcohol, was detected in the serum of patients 30 minutes post inhalation after a single dose of 110 mg or 220 mg of perillyl alcohol and lasted for 3 hours.

ELIGIBILITY:
Inclusion Criteria

Patient must:

1. Have histologically confirmed WHO Grade II or III meningioma that is residual, progressive or recurrent following at least minimally safe resection and radiation therapy. Metastatic meningiomas are allowed.

   1. Residual disease is defined as residual measurable disease (without a requirement for progression). Residual measurable disease is defined by bidimensionally measurable lesions with clearly defined margins by MRI scan(s) with a minimum diameter of 10mm in both dimensions.
   2. Progressive disease is defined as an increase in size of the measurable primary lesion on imaging by 25% or more (bidirectional area). The change must occur between scans separated by no more than 24 months.
   3. Recurrent disease is defined as new evidence of measurable disease following complete resection (10mm in both dimensions).
2. Be on a stable or decreasing dose of steroids for at least five days prior to the date of informed consent.
3. Participants must have failed maximal safe resection and radiation therapy.
4. There is no limit on the number of prior surgeries, radiation therapy, radiosurgery treatments or systemically administered therapeutic agents, however, these treatment(s) must comply with the following:

   1. There is no limit on the number of prior therapies.
   2. Prior medical therapy is allowed but is not required.
   3. No chemotherapy, other investigational agents within 14 days of study treatment.
   4. For prior systemic agents, participants must be at least 4 weeks (or 5 half-lives, whichever is shorter) from other prior cytotoxic chemotherapy (6 weeks from nitrosoureas/alkylating agents) or biologic therapies.
   5. No other concurrent receipt of investigational agents or other meningioma-directed therapy (chemotherapy, radiation) while on study.
   6. Patients may have been treated with standard external beam radiation or radiosurgery in any combination; however an interval of ≥12 weeks (84 days) must have elapsed from the completion of the radiation therapy to the initiation of study therapy unless there is histopathologic confirmation of recurrent tumor or there is new enhancing tumor outside the radiation field (beyond the high dose region or the 80% isodose line). In addition, there must be subsequent evidence of tumor progression after completion of radiation therapy;
   7. An interval of ≥ 28 days and full recovery (no ongoing safety issues) from surgical resection is required;
   8. Meningiomas that have resulted from prior radiation therapy are allowed.
   9. There must be an interval of ≥ 7 days from stereotactic biopsy; and
5. Participants must have recovered to grade ≤1 or pretreatment baseline from clinically significant adverse events related to prior therapy (exclusions include, but are not limited to alopecia, laboratory values listed per inclusion criteria and lymphopenia)
6. Patient must be ≥ 12 years of age.
7. Patient must have an ECOG performance status of 0-2 or KPS ≥ 60.
8. Patient must have an expected survival of at least three months.
9. Patient must be willing to provide blood sample for pharmacokinetic study (to assess proper administration of NEO100).
10. Patient must have adequate organ and marrow function as defined below:
11. White blood cell (WBC) ≥2000/microliter
12. Absolute neutrophil count (ANC) ≥ 1,500/microliter
13. Platelets ≥ 100,000/microliter
14. Hemoglobin ≥9 gm/dl
15. AST (SGOT)/ALT (SPGT) ≤ 2.5 × laboratory upper limit of normal (ULN)
16. Serum creatinine ≤ 1.5 x laboratory upper limit of normal (ULN) or
17. Creatinine clearance (meas or calc) ≥60mL/min for participants with creatinine levels >1.5x laboratory upper limit of normal (ULN)
18. Total serum bilirubin ≤ 1.5 x laboratory upper limit of normal (ULN) except participants with Gilbert's Syndrome who can have a total serum bilirubin of <5 x laboratory upper limit of normal (ULN)
19. MRI (or CT if MRI contraindicated) within 14 days prior to start of study drug. Corticosteroid dose must be stable or decreasing for at least 5 days prior to the scan. If steroids are added or the steroid dose is increased between the date of the screening scan and the start of treatment, a new baseline scan is required.
20. Female patients of child-bearing potential and male patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for 30 days prior to the first administration of study drug, for the duration of study participation, and for 90 days following completion of therapy. Should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
21. A female of child-bearing potential is any woman (regardless of sexual orientation, not having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    1. Has not undergone a hysterectomy or bilateral oophorectomy; or
    2. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
22. A negative serum pregnancy test will be required of all female patients of child-bearing potential within seven days prior to initiating study drug.
23. A serum pregnancy test will be repeated immediately if pregnancy is suspected.
24. Women must not be breastfeeding.
25. Patient must have the ability to understand, and the willingness comply with scheduled visits, treatment schedule, laboratory testing and other requirements of the study as confirmed by signing a written informed consent document.

Exclusion Criteria

1. Patients who have had chemotherapy, targeted small molecule therapy or study therapy within 14 days (or 5 half-lives, whichever is shorter) of study treatment.
2. Patient has completed chemo-radiation within the last 84 days prior to the first administration of study drug, unless new contrast enhancement is outside of radiation field, or there is tissue proven recurrence or progression.
3. Patient has had surgery within seven days prior to the date of informed consent.
4. Patient has had cytotoxic chemotherapy within 4 weeks (or 5 half-lives, whichever is shorter), nitrosoureas/alkylating agents within 6 weeks or biologic therapies.
5. Prior treatment with interstitial brachytherapy within 6 months of start of study therapy.
6. Current or planned participation in a clinical trial of an investigational agent or using an investigational medical device.
7. The patient's disease is primarily localized to the brainstem or spinal cord;
8. Patient has not recovered from adverse events due to chemotherapy, immunotherapy, or radiation therapy.
9. Patient has had prior treatment with perillyl alcohol.
10. Patient has a history of allergic reactions attributed to perillyl alcohol.
11. Patient has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
12. Patient must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
13. Patient has a history of new diagnosis or treatment of cancer other than high-grade meningioma within five years prior to the date of informed consent, except for basal cell carcinoma or squamous cell carcinoma of the skin.
14. Leptomeningeal involvement of the patient's tumor.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival as six months (PFS6). | 6 months
  Progression free survival

SECONDARY OUTCOMES:
Objective Tumor response to NEO100 as determined by RANO criteria | 6 months
Overall survival | 12 months
Perillic acid measurement | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Tom Chen, MD, PhD, Study Chair — NeOnc Technologies; Josh Neman, Study Director — NeOnc Technologies Holdings, Inc.
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided